CLINICAL TRIAL: NCT06574711
Title: Evaluation of the Effect of Consuming Yogurts Fortified With Dietary Sources of Vitamin E and Omega-3 on Classical Biomarkers of Cardiovascular Disease and Blood Levels of Vitamin E.
Brief Title: Functional Yogurt Consumption and Its Effects on the Lipid Profile of Healthy Subjects
Acronym: FYOPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Javeriana (Other)
Collaborators: Universidad Nacional de Colombia (Other)
Responsible Party: Principal Investigator, Ruby Alejandra Villamil, Principal investigator, Pontificia Universidad Javeriana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20415
Record Dates: First submitted 2024-08-14; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases; Apolipoproteins; Food Preferences; Low-density-lipoprotein-type; HDL; Triglycerides; Functional Food
Keywords: PUFA; cardiovascular risk; lipid profile; healthy volunteers; yogurt; sacha inchi oil; interspecific hybrid palm oil
MeSH Terms: conditions — Cardiovascular Diseases; Food Preferences

STUDY DESIGN:
Intervention Model Description: A pilot randomized; double-blind, parallel-controlled pragmatic trial was performed
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Forty-seven subjects were randomized and assigned to one of the three intervention groups supplemented daily with 200g of: Sacha Inchi Oil (SIO)-containing yogurt (Group-A), Hybrid palm oil (HPO)-containing yogurt (Group-B), and plain yogurt (Group-C).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control yogurt (Placebo Comparator): Participants consumed a 200 g bottle of plain Yogurt with 3.5% unreplaced fat orally, daily, for 90 days
  Interventions: Other: Control yogurt
- Sacha inchi oil yogurt (Experimental): Participants consumed a 200 g bottle of Yogurt with 3.5% replacement of dairy fat for Sacha inchi oil, orally, daily, for 90 days
  Interventions: Other: Sacha inchi oil yogurt
- Hybrid palm oil yogurt (Experimental): Participants consumed a 200 g bottle of Yogurt with 3.5% replacement of dairy fat for Hybrid Palm Oil, daily, for 90 days
  Interventions: Other: Hybrid palm oil yogurt

INTERVENTIONS:
Other: Sacha inchi oil yogurt — Sacha inchi oil was incorporated into a nonfat yogurt acting as a source of linolenic acid
  Arms: Sacha inchi oil yogurt
Other: Hybrid palm oil yogurt — Interspecific hybrid palm oil was incorporated into a nonfat yogurt as a source of bioactive compounds
  Arms: Hybrid palm oil yogurt
Other: Control yogurt — Conventional full-fat yogurt
  Arms: Control yogurt

SUMMARY:
The purpose of this study was to assess the effect of the daily intake of yogurts enhanced with Sacha Inchi oil and hybrid palm tree oil on human plasma lipids related to cardiovascular risk factors

DETAILED DESCRIPTION:
After being recruited and signing a written informed consent about the study and potential risks, the participants were randomized and assigned in a double-blind manner to one of three intervention groups (control yogurt, sacha inchi oil yogurt, or hybrid palm tree oil yogurt; consumption 1 bottle of 200ml per day for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Normal total cholesterol (≤200mg/dl) levels
* Have a yogurt consumption habit of at least three times a week
* Maximum level of moderate physical activity
* Body mass index (BMI) of ≤29.9kg/m2
* Serum triacylglycerols below 400mg/dl

Exclusion Criteria:

* Presence of chronic disease (Arterial hypertension, Diabetes Mellitus, among others)
* A history of illicit drug use and/or chronic alcohol use, active smoking
* A well-established allergy to red palm olein and/or milk and its derivatives
* Consumption of nutritional supplements (antioxidants, omega 3, fiber, phytosterols)
* Pregnancy or lactation
* Having menopause
* High consumption of nuts, flaxseed, chia, and sesame seeds

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Change in plasma levels of total cholesterol | Baseline, 1 month, 2 months and 3 months
  Measure in plasma (mmol/l)
Change in plasma levels of LDL-cholesterol | Baseline, 1 month, 2 months and 3 months
  Measure in plasma (mmol/l)
Change in plasma levels of HDL-cholesterol | Baseline, 1 month, 2 months and 3 months
  Measure in plasma (mmol/l)
Change in plasma levels of triacylglycerols | Baseline, 1 month, 2 months and 3 months
  Measure in plasma (mmol/l)
Change in plasma levels of Apolipoprotein A1 (ApoA1) | Baseline, 1 month, 2 months and 3 months
  Measure in plasma (g/l)
Change in plasma levels of Apolipoprotein B (ApoB) | Baseline, 1 month, 2 months and 3 months
  Measure in plasma (g/l)
ApoB/ApoA1 ratio | Baseline, 1 month, 2 months and 3 months
  prognostic predictor of a 10 year cardiovascular event

CONTACTS AND LOCATIONS:
Overall Officials: Lilia Y Cortés, PhD, Study Director — Pontificia Universidad Javeriana
Locations (1):
- Pontificia Universidad Javeriana, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No
Due to the informed consent, no individual data can be shared; however, the results will be shared in a scientific publication

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT06574711/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT06574711/ICF_001.pdf